CLINICAL TRIAL: NCT06752369
Title: Adapting Single Sessions Interventions for Type 1 Diabetes (ASSISTED): Integrated Pediatric Care to Reduce Depression and HbA1c
Brief Title: Adapting Single Sessions Interventions for Type 1 Diabetes
Acronym: ASSISTED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Health System (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Alexandra Monzon, Assistant Research Scientist, Nemours Children's Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23DK139431 (NIH); K23DK139431 (NIH)
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: type 1 diabetes; adolescents; depression
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T1D-specific depression SSI (Experimental): Single session depression intervention adapted for youth with T1D. The T1D-specific depression SSI will include 1) psychoeducation about depression, including how behavior shapes feelings and thoughts, 2) a values assessment, where youth will identify key areas (i.e., family relationships, friendships, school, or hobbies) from which they draw (or once drew) enjoyment and meaning, and 3) the creation of an activity action plan, wherein youth identify (from pre-generated lists) and personalize (in guided exercises) three activities to target for change.
  Interventions: Behavioral: T1D-specific depression SSI
- T1D Education (Placebo Comparator): Educational material about T1D
  Interventions: Behavioral: T1D Educational

INTERVENTIONS:
Behavioral: T1D-specific depression SSI — The T1D-specific depression SSI will include 1) psychoeducation about depression, including how behavior shapes feelings and thoughts, 2) a values assessment, where youth will identify key areas (i.e., family relationships, friendships, school, or hobbies) from which they draw (or once drew) enjoyment and meaning, and 3) the creation of an activity action plan, wherein youth identify (from pre-generated lists) and personalize (in guided exercises) three activities to target for change.
  Arms: T1D-specific depression SSI
Behavioral: T1D Educational — T1D Educational Material
  Arms: T1D Education

SUMMARY:
The goal of this clinical trial is to learn if implementing a single-session depression intervention for youth with type 1 diabetes (T1D) is feasible and acceptable to patients. can help improve mood and health outcomes. It will also learn about the initial efficacy of the intervention. The main questions it aims to answer are:

1. Is a single-session depression intervention for youth with T1D feasible to recruit and implement?
2. Is a single-session depression intervention for youth with T1D acceptable to patients (i.e., do they find it helpful)?
3. Does a single-session depression intervention for youth with T1D lead to improvements in low mood?

Researchers will compare a single-session depression intervention for youth with to a education control to see if a single-session depression intervention works to improve depressive symptoms.

Participants will:

* Participate in a single-session depression intervention
* Complete questionnaires and provide a sample for A1c at a baseline, 3-month, and 6-month visit
* Complete daily questionnaires once a day for two weeks before and after the single-session depression intervention

ELIGIBILITY:
Inclusion Criteria:

* Child or adolescent age between 11-18 years, inclusive
* Physician confirmed T1D diagnosis of at least 6 months duration prior to study enrollment
* Positive depression screening score of >5 on the PHQ-9 in the last year
* Not currently engaged in outpatient mental healthcare
* English fluency

Exclusion Criteria:

* Another systemic chronic medical illness except for celiac disease, autoimmune thyroiditis, microalbuminuria, hypertension, or well-managed asthma
* Any score of 1, 2, or 3 on item 9 (indicating suicidal ideation) of the PHQ-9 in the last year.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | 0, 3-months, and 6-months
  Proxy measure of glycemic level. HbA1c is the average blood glucose level over 3-4 months. We will use fingerstick blood samples and a valid mail-in dried blood spot kit to measure participant HbA1c levels at a central laboratory
Patient Health Questionnaire for Adolescents (PHQ-9) | 0, 3-months, and 6-months
  The PHQ-9 is a well-validated and reliable measure that assesses the occurrence of nine possible depressive symptoms over the previous two weeks. Higher scores indicate greater depressive symptoms. A cut-off score of >5 will be used to characterize elevated depressive symptoms
Positive and Negative Affect Schedule (PANAS) | 7 days before and 7 days after SSI
  The PANAS is a 20-item measure that assesses different feelings and emotions. Items are grouped into the two subscales with 10 items each: positive affect and negative affect, with higher scores on the Positive Affect subscale indicating greater intensity of positive emotions, and higher scores on the Negative Affect subscale indicating greater intensity of negative emotions.
Mood and Feelings Questionnaire (MFQ) | 7 days before and 7 days after SSI
  The MFQ is a 13-item measure that assesses depressed mood in youth. Higher scores indicate higher depressed mood.
Feasibility of T1D-specific Depression SSI | Baseline and 3-months
  We will determine feasibility by calculating study enrollment rates for the Aim 2 pilot trial. We will also assess the feasibility of the type 1 diabetes (T1D)-specific depression single-session intervention (SSI) in the qualitative interviews
Acceptability of Healthcare Interventions Questionnaire | immediately after SSI completion
  The Acceptability of Healthcare Interventions Questionnaire is an 8-item measure that assesses the acceptability of healthcare interventions. Respondents rate each question on a scale of
  1 (strongly disagree) to 5 (strongly agree), with higher scores indicating greater intervention acceptability.

SECONDARY OUTCOMES:
Problem Areas in Diabetes- Teen (PAID-T) | 0, 3-months, and 6-months
  The PAID-T is a 26-item measure that assesses diabetes-specific emotional distress in adolescents with T1D. Adolescents rate how much each item applies to them on a 6-point Likert scale from 1 (Not a Problem) to 6 (Serious Problem), with higher scores indicating greater distress.
Diabetes Family Conflict Scale- Revised (DFCS-R) | 0, 3-months, and 6-months
  The DFCS-R is a 19-item measure that evaluates conflict between youth and their caregivers surrounding direct and indirect diabetes management tasks. Adolescents will rate how often they argue with their parents on a 3-point Likert scale ranging from 1 (Never Argue) to 3 (Always Argue), with higher scores indicating more parent-child conflict.
Diabetes Strengths and Resilience Measure for Adolescents (DSTAR-Teen) | 0, 3-months, 6-months
  The DSTAR-teen is a 12-item measure that assesses adaptive behaviors and attitudes about diabetes in adolescents with T1D. Adolescents rate how often each item occurs for them on a 5 -point Likert scale from 1 (Never) to 5 (Almost Always), with higher scores indicating greater strength and resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Hospital - FL, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided